CLINICAL TRIAL: NCT02683863
Title: An Open Label Study of the Pharmacokinetics of DMF and the Effects of DMF on Exploratory Biomarkers in Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: Pharmacokinetics of DMF and the Effects of DMF on Exploratory Biomarkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Multiple Sclerosis Center of Northeastern New York (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG12-001
Record Dates: First submitted 2016-01-14; First posted 2016-02-17 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Other): There will be 4 CSF sampling groups at the Week 6 visit for PK assessment:
  1. Four subject for CSF samples 3 hours after dosing
  Interventions: Drug: BG00012 (DMF) (Tecfidera®.)
- Group 2 (Other): 2. Four subjects for CSF samples 5 hours after dosing
  Interventions: Drug: BG00012 (DMF) (Tecfidera®.)
- Group 3 (Other): 3. Four subjects for CSF samples 7 hours after dosing
  Interventions: Drug: BG00012 (DMF) (Tecfidera®.)
- Group 4 (Other): 4. Four subjects for predose CSF samples
  Interventions: Drug: BG00012 (DMF) (Tecfidera®.)

INTERVENTIONS:
Drug: BG00012 (DMF) (Tecfidera®.) — Subjects will take DMF 120 mg BID for the first 4 weeks of treatment followed by DMF 240 mg BID for 24 weeks.

SUMMARY:
The purpose of this study is to explore whether DMF (Dimethyl Fumarate) or MMF (monomethyl fumarate) its main bioactive metabolite, is capable of entering the central nervous system in SPMS patients that are being treated with Tecfidera®. PK samples (pharmacokinetics - or the amount of study drug in blood) will be tested to compare with PK samples, the amount of study drug, in spinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria (MS Population):

To be eligible to participate in this study, candidates must meet the following eligibility criteria at screening, or at the timepoint specified in the individual eligibility criterion listed:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local patient privacy regulations. Subjects must provide separate informed consent to participate in this CSF study.
2. Aged 25 to 65 years-old, inclusive, at the time of informed consent.
3. Male of female subject with a confirmed diagnosis of SPMS.
4. EDSS score between 3 and 7, inclusive, at screening.
5. Weight should be between 130 and 200 lb.

Exclusion Criteria (MS Population)

* Candidates will be excluded from study entry if any of the following exclusion criteria exist at screening, or at the timepoint specified in the individual criterion listed:

  1. Unable or unwilling to provide informed consent. (Subjects must provide separate informed consent for this study.)
  2. A MS relapse, as determined by the Investigator, which occurred within 90 days prior to screening, or the subject has not stabilized from a previous relapse prior to screening.
  3. Any contraindication to having a brain magnetic resonance imaging (MRI) (e.g., pacemaker, MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed) or contraindication for administration of gadolinium-contrast agent.
  4. Clinically significant brain MRI finding other than those related to MS, as judged by the Investigator, at screening.
  5. Any contraindications to having a LP (e.g., aspirin greater than 325 mg/day, warfarin, clopidrogel, decreased platelet count, prolonged PT or PTT more than 1 ½ over normal) as determined by history and Investigator decision.
  6. Evidence of history of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, ulcerative colitis, diabetes mellitus) with the exception of MS.
  7. Any sign of chronic active infection, requiring antibiotic treatment (refer to Exclusion 23) (e.g., urinary tract infection, bronchitis, hepatitis, and tuberculosis) except for those requiring topical medication for treatment (e.g., athletes foot), or screening laboratory evidence consistent with a significant chronic active acute infection requiring systemic treatment.
  8. Pregnant; or breastfeeding females; or males of fathering potential or females of childbearing potential who are unwilling or unable to use an effective method of contraception as outlined in this protocol (Section 12.5) for the duration of the study and for at least 28 days after the last dose of DMF use in this protocol. For females of childbearing potential, a positive pregnancy test at any time within the protocol.
  9. Known positive human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody tests indicative of present or prior infection.
  10. Any abnormal hematology values or clinical chemistry values judged by the Investigator or Sponsor as clinically significant, including white blood cell count (WBC) 3500/mm3, or absolute lymphocyte count lower limit of normal.
  11. Positive Quantiferon-Tuberculosis Gold In-Tube test (QFT-GIT) at screening or known history of active tuberculosis not adequately treated.
  12. Any malignancy within 5 years, except for basal or squamous cell skin lesions which have been surgically excised, with no evidence of metastasis.
  13. Any clinical, CSF, or MRI evidence for progressive multifocal leukoencephalopathy, from historical MRI.
  14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
  15. Subjects participating in or expecting to participate in other interventional clinical trials, except those participating in Study US-BGT-US-10766 at the same site.
  16. History of drug or alcohol abuse (as defined by the Investigator) within 2 years prior to screening.

      Exclusion Criteria Related to Medication
  17. Previous exposure to DMF for disease management at any time in the past.
  18. History of severe allergic or anaphylactic reactions or known drug hypersensitivity to fumaric acid or fumaric acid esters.
  19. Treatment with methylprednisolone or other systemic corticosteroid for MS relapse or otherwise within 30 days prior to Day 1 of study treatment.
  20. Treatment with MS disease modifying therapies as follows:

      Beta interferons (interferon beta-1a [Avonex® or Rebif®] or interferon beta-1b [Betaseron®], or glatiramer acetate [Copaxone®] within 6 weeks prior to Baseline.

      Fingolimod (Gilenya®), teriflunomide (Aubagio®) within 6 months prior to Baseline, except teriflunomide washout with accelerated elimination and verification of zero serum levels of teriflunomide prior Baseline.

      Natalizumab (Tysabri®) within 6 months prior to Screening OR 1 month prior to screening if subject has a positive Nabs (neutralizing antibodies) to Tysabri® Treatment within the past 5 years or current treatment with any of the following agents: cyclosporine, cladribine, agents that are immunosuppressive (e.g., entanercept), murine protein, T-cell vaccination), or stem cell transplantation prior to Screening.

      Treatment within the past 2 years with rituximab, IVIG, or mycophenolate
  21. Receipt of any non-live vaccine within the previous 14 days or live vaccine within 30 days prior to first dose of study treatment.
  22. Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study treatment, whichever is longer.
  23. Use of antibiotics for any reason within 3 months of Screening. Inclusion Criteria (for Normal Control Volunteers Only)

To be eligible to participate in this study, normal control candidates must meet the following eligibility criteria at screening:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local patient privacy regulations. Subjects must provide separate informed consent to participate in this CSF study.
2. Male or female, aged 25 to 65 years-old, inclusive, at the time of informed consent.
3. Weight should be between 130 and 200 lb. Exclusion Criteria (for Normal Control Volunteers Only)

Normal control candidates will be excluded from study entry if any of the following exclusion criteria exist at screening, or at the timepoint specified in the individual criterion listed:

1. Unable or unwilling to provide informed consent. (Subjects must provide separate informed consent for this study.)
2. Any contraindications to having a LP (e.g., aspirin greater than 325 mg/day, warfarin, clopidrogel, decreased platelet count, prolonged PT or PTT more than 1 ½ over normal) as determined by history and Investigator decision.
3. Evidence of history of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, ulcerative colitis, diabetes mellitus) with the exception of MS.
4. Any sign of chronic active infection, requiring antibiotic treatment (refer to Exclusion 23) (e.g., urinary tract infection, bronchitis, hepatitis, and tuberculosis) except for those requiring topical medication for treatment (e.g., athletes foot), or screening laboratory evidence consistent with a significant chronic active acute infection requiring systemic treatment.
5. Pregnant; or breastfeeding females; or males of fathering potential or females of childbearing potential who are unwilling or unable to use an effective method of contraception as outlined in this protocol (Section 12.5) for the duration of the study and for at least 28 days after the last dose of DMF use in this protocol. For females of childbearing potential, a positive pregnancy test at any time within the protocol.
6. Known positive human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody tests indicative of present or prior infection.
7. Any abnormal hematology values or clinical chemistry values judged by the Investigator or Sponsor as clinically significant, including white blood cell count (WBC) 3500/mm3, or absolute lymphocyte count lower limit of normal.
8. Positive Quantiferon-Tuberculosis Gold In-Tube test (QFT-GIT) at screening or known history of active tuberculosis not adequately treated.
9. Any malignancy within 5 years, except for basal or squamous cell skin lesions which have been surgically excised, with no evidence of metastasis.
10. Any clinical, CSF, or MRI evidence for progressive multifocal leukoencephalopathy, from historical MRI.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
12. Subjects participating in or expecting to participate in other interventional clinical trials, except those participating in Study US-BGT-US-10766 at the same site.
13. History of drug or alcohol abuse (as defined by the Investigator) within 2 years prior to screening.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to investigate the PK (drug level) of DMF(study drug) in CSF with SPMS. | post-DMF treatment in Week 6
  Concentration of DMF in CSF predose and at 3, 5, 7 hours post DMF treatment in week 6.
The primary objective of the study is to investigate the PK (drug level) of DMF(study drug) in plasma in subjects with SPMS. | treatment in week 6
  Concentration of DMF in plasma predose and at 2,3,5,6, 7 and 8 hours post-DMF treatment at Week 6
The primary objective of the study is to investigate the PK (drug level) of MMF(the primary metabolite of study drug) in CSF with SPMS. | treatment in week 6
  Concentration of MMF in CSF predose and at 3, 5, 7 hours post DMF treatment in week 6.
The primary objective of the study is to investigate the PK (drug level) of MMF( the primary metabolite of study drug) in plasma in subjects with SPMS. | treatment in week 6
  Concentration of MMF in plasma predose and at 2,3,5,6, 7 and 8 hours post-DMF treatment at Week 6
The primary objective of the study is to investigate the PK (drug level) of DMF conjugate (study drug) in CSF with SPMS. | treatment in week 6
  Concentration of DMF conjugate in CSF predose and at 3, 5, 7 hours post DMF treatment in week 6.
The primary objective of the study is to investigate the PK (drug level) of DMF conjugate (study drug) in plasma in subjects with SPMS. | treatment in week 6
  Concentration of DMF conjugate in plasma predose and at 2,3,5,6, 7 and 8 hours post-DMF treatment at Week 6
The primary objective of the study is to investigate the PK (drug level) of MMF (the primary metabolite of study drug) conjugate in CSF with SPMS. | treatment in week 6
  Concentration of MMF conjugate in CSF predose and at 3, 5, 7 hours post DMF treatment in week 6.
The primary objective of the study is to investigate the PK (drug level) of MMF( the primary metabolite of study drug) conjugate in plasma in subjects with SPMS. | treatment in week 6
  Concentration of MMF conjugate in plasma predose and at 2,3,5,6, 7 and 8 hours post-DMF treatment at Week 6

SECONDARY OUTCOMES:
A secondary objective is to assess the effects of DMF on PD biomarkers downstream of Nrf2 in the CSF of subjects with SPMS. | at 28 weeks
  PD biomarkers downstream of Nrf2, such as NAD(P)H hydrogenase [quinone 1], heme oxygenase-1, and aldo-keto reductase family 1 member B8 that have not been evaluated in CNS.
A secondary objective is to assess the effects of DMF on biomarkers of inflammation in the CSF of subjects with SPMS. | at 28 weeks
  Biomarkers of inflammation (e.g., osteopontin, B cell activating factor, chemokines, and matrix metalloproteinase 9), which may reflect pathogenesis in SPMS.
A secondary objective is to assess the effects of DMF on biomarkers of neuroaxonal damage in the CSF of subjects with SPMS. | at 28 weeks
  Biomarkers of neuroaxonal damage (e.g., neurofilament, myelin basic protein, glial fibrillary acidic protein, and neural cell adhesion molecule), which may reflect pathogenesis in SPMS.
A secondary objective is to assess the effects of DMF on biomarkers of oxidative stress in the CSF of subjects with SPMS. | at 28 weeks
  Biomarkers of oxidative stress (e.g., myeloperoxidase, 8-Oxo-2'-deoxyguanosine and RNA biomarkers), which may reflect pathogenesis in SPMS
A secondary objective is to assess the effects of DMF on myelin lipid biomarkers in the CSF of subjects with SPMS. | at 28 weeks
  Myelin lipid biomarkers (e.g., cholesterol, galactoceramide, sulfatides, and sphingomyelin), which may correlate with disability progression in MS patients.
A secondary objective is to assess the effects of DMF on pharmacogenomic biomarkers in the CSF of subjects with SPMS. | at 28 weeks
  Pharmacogenomic biomarkers: DNA analysis from blood samples.
A secondary objective is to assess the effects of DMF on RNA samples from CSF cellular pellet for transcriptionomics in the CSF of subjects with SPMS. | at 28 weeks
  RNA samples from CSF cellular pellet for transcriptionomics.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Edwards, M.D, Principal Investigator — MS Center of Northeastern NY
Locations (1):
- Multiple Sclerosis Center of Northeastern New York, Latham, New York, United States

REFERENCES:
- [Background] Lassmann H, van Horssen J, Mahad D. Progressive multiple sclerosis: pathology and pathogenesis. Nat Rev Neurol. 2012 Nov 5;8(11):647-56. doi: 10.1038/nrneurol.2012.168. Epub 2012 Sep 25. PMID 23007702
- [Background] Frischer JM, Bramow S, Dal-Bianco A, Lucchinetti CF, Rauschka H, Schmidbauer M, Laursen H, Sorensen PS, Lassmann H. The relation between inflammation and neurodegeneration in multiple sclerosis brains. Brain. 2009 May;132(Pt 5):1175-89. doi: 10.1093/brain/awp070. Epub 2009 Mar 31. PMID 19339255
- [Background] Kutzelnigg A, Lucchinetti CF, Stadelmann C, Bruck W, Rauschka H, Bergmann M, Schmidbauer M, Parisi JE, Lassmann H. Cortical demyelination and diffuse white matter injury in multiple sclerosis. Brain. 2005 Nov;128(Pt 11):2705-12. doi: 10.1093/brain/awh641. Epub 2005 Oct 17. PMID 16230320
- [Background] Lassmann H. New concepts on progressive multiple sclerosis. Curr Neurol Neurosci Rep. 2007 May;7(3):239-44. doi: 10.1007/s11910-007-0036-0. PMID 17488590
- [Background] Calkins MJ, Johnson DA, Townsend JA, Vargas MR, Dowell JA, Williamson TP, Kraft AD, Lee JM, Li J, Johnson JA. The Nrf2/ARE pathway as a potential therapeutic target in neurodegenerative disease. Antioxid Redox Signal. 2009 Mar;11(3):497-508. doi: 10.1089/ars.2008.2242. PMID 18717629
- [Background] Linker RA, Lee DH, Ryan S, van Dam AM, Conrad R, Bista P, Zeng W, Hronowsky X, Buko A, Chollate S, Ellrichmann G, Bruck W, Dawson K, Goelz S, Wiese S, Scannevin RH, Lukashev M, Gold R. Fumaric acid esters exert neuroprotective effects in neuroinflammation via activation of the Nrf2 antioxidant pathway. Brain. 2011 Mar;134(Pt 3):678-92. doi: 10.1093/brain/awq386. PMID 21354971
- [Background] Scannevin RH, Chollate S, Jung MY, Shackett M, Patel H, Bista P, Zeng W, Ryan S, Yamamoto M, Lukashev M, Rhodes KJ. Fumarates promote cytoprotection of central nervous system cells against oxidative stress via the nuclear factor (erythroid-derived 2)-like 2 pathway. J Pharmacol Exp Ther. 2012 Apr;341(1):274-84. doi: 10.1124/jpet.111.190132. Epub 2012 Jan 20. PMID 22267202
- [Background] Ellrichmann G, Petrasch-Parwez E, Lee DH, Reick C, Arning L, Saft C, Gold R, Linker RA. Efficacy of fumaric acid esters in the R6/2 and YAC128 models of Huntington's disease. PLoS One. 2011 Jan 31;6(1):e16172. doi: 10.1371/journal.pone.0016172. PMID 21297955
- [Background] Ghoreschi K, Bruck J, Kellerer C, Deng C, Peng H, Rothfuss O, Hussain RZ, Gocke AR, Respa A, Glocova I, Valtcheva N, Alexander E, Feil S, Feil R, Schulze-Osthoff K, Rupec RA, Lovett-Racke AE, Dringen R, Racke MK, Rocken M. Fumarates improve psoriasis and multiple sclerosis by inducing type II dendritic cells. J Exp Med. 2011 Oct 24;208(11):2291-303. doi: 10.1084/jem.20100977. Epub 2011 Oct 10. PMID 21987655
- [Background] Gold R, Kappos L, Arnold DL, Bar-Or A, Giovannoni G, Selmaj K, Tornatore C, Sweetser MT, Yang M, Sheikh SI, Dawson KT; DEFINE Study Investigators. Placebo-controlled phase 3 study of oral BG-12 for relapsing multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1098-107. doi: 10.1056/NEJMoa1114287. PMID 22992073
- [Background] Fox RJ, Miller DH, Phillips JT, Hutchinson M, Havrdova E, Kita M, Yang M, Raghupathi K, Novas M, Sweetser MT, Viglietta V, Dawson KT; CONFIRM Study Investigators. Placebo-controlled phase 3 study of oral BG-12 or glatiramer in multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1087-97. doi: 10.1056/NEJMoa1206328. PMID 22992072
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061
- [Background] Comi G. Disease-modifying treatments for progressive multiple sclerosis. Mult Scler. 2013 Oct;19(11):1428-36. doi: 10.1177/1352458513502572. PMID 24062415